CLINICAL TRIAL: NCT00999076
Title: Rapid Identification of Mycobacteria in Acid-fast Bacilli Smear-positive Respiratory Specimens
Status: Terminated | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won-Jung Koh, Associate Professor, Samsung Medical Center
Other Study IDs: 2009-09-004
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Atypical Mycobacteria; Mycobacterium Infections
MeSH Terms: conditions — Mycobacterium Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum with positive AFB smear
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sputum with positive AFB smear

SUMMARY:
The aim of the study is to evaluate the polymerase chain reaction (PCR)-Reverse Blot Hybridization Assay (REBA) for identification of nontuberculous mycobacteria (NTM) species in acid-fast bacilli (AFB) smear-positive respiratory specimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AFB-smear positive sputum

Exclusion Criteria:

* Non-applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with AFB-smear positive sputum
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Results of REBA for identification of NTM species | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Won-Jung Koh, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea